CLINICAL TRIAL: NCT00483821
Title: A Retrospective Analysis of Neck Dissection Following Complete Response to Chemoradiation in HNSCC
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine; Director, Cancer Supportive Care Program; Director, Head and Neck Research Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC HN 0435; VU-VICC-HN-0435; VU-VICC-IRB-040428
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage I verrucous carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; stage I verrucous carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: medical chart review — medical chart review

SUMMARY:
RATIONALE: Gathering disease-related information from medical charts of patients with primary head and neck cancer who have undergone neck dissection after complete response to chemotherapy and radiation therapy may help doctors learn more about the disease and find better methods of treatment.

PURPOSE: This clinical trial is evaluating the medical charts of patients with primary head and neck cancer who have undergone neck dissection after complete response to chemotherapy and radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Perform a retrospective analysis, by medical chart review, of patients with primary squamous cell carcinoma of the head and neck who underwent neck dissection following complete response to chemoradiotherapy.
* Determine whether the role of a post-chemoradiotherapy neck dissection affects the outcome of the patient's disease, in terms of overall survival, disease-free survival, and recurrence rates.

OUTLINE: This is a pilot, retrospective study.

Patients who have undergone neck dissection after achieving a complete clinical and radiological response to chemoradiotherapy are compared to patients who did not. Data are gathered by medical chart review.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary squamous cell carcinoma of the head and neck at any of the following sites:

  * Oral cavity
  * Oropharynx
  * Hypopharynx
  * Larynx
* Complete response achieved after treatment with chemoradiotherapy

Exclusion Criteria:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with the diagnosis of primary squamous cell carcinoma of the head and neck at any of the following sites:
  * Oral cavity
  * Oropharynx
  * Hypopharynx
  * Larynx
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2004-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | off-study date

SECONDARY OUTCOMES:
Disease-free survival | off-study date
Recurrence rate | off-study date

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee